CLINICAL TRIAL: NCT04179175
Title: A Multicenter, Double-blind, Randomized Withdrawal Extension Study of Subcutaneous Secukinumab to Demonstrate Long-term Efficacy, Safety and Tolerability in Subjects With Moderate to Severe Hidradenitis Suppurativa
Brief Title: Extension Study to Assess Effects of Non-interrupted Versus Interrupted and Long Term Treatment of Two Dose Regimes of Secukinumab in Subjects With Hidradenitis Suppurativa
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAIN457M2301E1; 2023-508956-20 (Registry Identifier: CTIS (EU) Number)
Record Dates: First submitted 2019-11-25; First posted 2019-11-27 (Actual); Results first posted 2024-06-21 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Hidradenitis Suppurativa
Keywords: acne inversa; Hidradenitis suppurativa (HS); maladie de Verneuil; inflammatory disease; AIN457; AIN457M; Secukinumab; Loss of Response (LOR); Hidradenitis Suppurativa Clinical Response (HiSCR); interleukin-17A (IL-17A)
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — secukinumab

STUDY DESIGN:
Intervention Model Description: Multicenter, double-blind, randomized withdrawal extension, parallel group study followed by an open-label, active-treatment period with two Secukinumab dose regimens in approximately 856 patients with moderate to severe hidradenitis suppurativa (HS)
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patients considered HiSCR responders will be randomized 2:1 to continue their current regimen or undergo withdrawal to placebo. HiScr non-responders will enter open label therapy with Secukinumab if desired
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- secukinumab 1 HiSCR Responder (Active Comparator): HiSCR responder at Week 52 in core trial, secukinumab 300mg every 2 weeks
  Interventions: Drug: secukinumab
- secukinumab 2 HiSCR Responder (Active Comparator): HiSCR responder at Week 52 in core trial, secukinumab 300mg every 4 weeks
  Interventions: Drug: secukinumab
- placebo 1 HiSCR Responder (Placebo Comparator): HiSCR responder at Week 52 in core trial, placebo to secukinumab 300mg every 2 weeks
  Interventions: Drug: secukinumab
- placebo 2 HiSCR Responder (Placebo Comparator): HiSCR responder at Week 52 in core trial, placebo to secukinumab 300 mg every 4 weeks
  Interventions: Drug: secukinumab
- HiSCR non-responders (Other): non-responder at Week 52 in core trial treatment; secukinumab 300mg every 2 weeks
  Interventions: Drug: secukinumab

INTERVENTIONS:
Drug: secukinumab — secukinumab 300mg every 2 weeks
  Other Names: AIN457
  Arms: HiSCR non-responders; placebo 1 HiSCR Responder; secukinumab 1 HiSCR Responder
Drug: secukinumab — secukinumab 300mg every 4 weeks
  Other Names: AIN457
  Arms: placebo 2 HiSCR Responder; secukinumab 2 HiSCR Responder

SUMMARY:
The purpose of this extension study is to evaluate maintenance of Hidradenitis Suppurativa Clinical Response (HiSCR response) in either continuous or interrupted therapy (using a randomized withdrawal period) of two dose regimens and to assess long-term efficacy, safety and tolerability of Secukinumab in subjects with moderate to severe hidradenitis suppurativa completing either of the 2 Phase III studies. This is an expanded access trial for the core trials CAIN457M2301 (NCT03713619) and CAIN457M2302 (NCT03713619).

DETAILED DESCRIPTION:
This is a multicenter extension study to both core Phase III studies CAIN457M2301 and CAIN457M2302 (Core studies). This study contains a randomized withdrawal design, double blinded and placebo controlled up to Week 104 or loss of response. The subjects with HiSCR response after 52 weeks of treatment in the "Core studies" will be randomized at 2:1 ratio to either continue on one of the two Secukinumab dosing regimens assigned in "Core studies" for another 52 weeks or will be placed on placebo. The primary endpoint is loss of response (LOR) assessed during the 52-week treatment duration (up to Week 104). Subjects who attained LOR will be transferred to open-label treatment to continue until the end of the study. Subjects on placebo who did not reach LOR up to Week 104 will be offered to continue in the open-label treatment or discontinue the study. Thus for subjects who were HiSCR responders at Week 52 of "Core studies", the open label treatment duration will vary and start either from the time of LOR or from Week 104 dose and last until Week 260 followed by 8 weeks of a post treatment follow-up period to week 268.

Subjects who were HiSCR non-responders at the end of "Core studies" will be offered to continue in open-label treatment until Week 260.

Subjects who prematurely discontinue the study, or who complete the study will enter a post-treatment follow up period (8 weeks) The primary objective is to evaluate maintenance of HiSCR response at Week 104 in either continuous or interrupted therapy compared to placebo. Secondary objectives are to assess the long-term safety and tolerability evaluated by adverse events, abnormal laboratory values and vital signs.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent must be obtained before any assessment is performed
* subject must have completed the study treatment period (52 weeks) in the core studies (AIN457M2301 or AIN457M2302) and had received secukinumab treatment during Treatment Period 2

Exclusion Criteria:

* protocol deviation in the core study which will prevent the meaningful analysis of the extension study
* ongoing or planned use of prohibited HS or non-HS treatment
* participation in the extension could expose the subject to an undue safety risk
* current sever progressive or uncontrolled disease which renders the subject unsuitable for the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 703 (Actual)
Dates: Start 2020-03-18 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2026-07-15 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (180):
- United States (29):
  - Northwest Arkansas Center, Rogers, Arkansas
  - MedDerm Associates, San Diego, California
  - University Clinical Trials, San Diego, California
  - Southern California Skin and Laser, Whittier, California
  - Florida Academic Centers Research and Education LLC, Coral Gables, Florida
  - University of MiamiHealth System, Miami, Florida
  - Olympian Clinical Research, Tampa, Florida
  - University Of South Florida, Tampa, Florida
  - Advanced Medical Research, Sandy Springs, Georgia
  - Endeavor Health, Glenview, Illinois
  - Dundee Dermatology, West Dundee, Illinois
  - Dawes Fretzin Clinical Rea Group, Indianapolis, Indiana
  - Tufts Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Med Center, Boston, Massachusetts
  - Minnesota Clinical Study Center, New Brighton, Minnesota
  - MediSearch Clinical Trials, Saint Joseph, Missouri
  - St Louis U Clinical Trials, St Louis, Missouri
  - WA Uni School Of Med, St Louis, Missouri
  - Skin Specialists PC, Omaha, Nebraska
  - Icahn School Of Med At Mount Sinai, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Wright State University, Fairborn, Ohio
  - UP Medical Center H System, Pittsburgh, Pennsylvania
  - Clinical Research Ctr of Carolinas, Charleston, South Carolina
  - Bellaire Dermatology Associates, Bellaire, Texas
  - MDRI Baylor University, Dallas, Texas
  - Austin Inst for Clinical Research, Pflugerville, Texas
  - Dr. Stephen Miller, MDPA, San Antonio, Texas
  - Virginia Clinical Research, Norfolk, Virginia
- Argentina (6):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, La Plata, Buenos Aires
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Caba
  - Novartis Investigative Site, Capital Federal
- Australia (3):
  - Novartis Investigative Site, Phillip, Australian Capital Territory
  - Novartis Investigative Site, Benowa, Queensland
  - Novartis Investigative Site, East Melbourne, Victoria
- Austria (2):
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Vienna
- Belgium (3):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Liège
- Bulgaria (3):
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Stara Zagora
- Canada (4):
  - Novartis Investigative Site, Barrie, Ontario
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Peterborough, Ontario
  - Novartis Investigative Site, Waterloo, Ontario
- Novartis Investigative Site, Barranquilla, Atlántico, Colombia
- Novartis Investigative Site, Zagreb, HRV, Croatia
- Czechia (4):
  - Novartis Investigative Site, Prague, Prague 1
  - Novartis Investigative Site, Jihlava
  - Novartis Investigative Site, Plzen Bory
  - Novartis Investigative Site, Ústí nad Labem
- France (17):
  - Novartis Investigative Site, Limoges, Haute Vienne
  - Novartis Investigative Site, Toulon, Val De Marne
  - Novartis Investigative Site, Antony
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Brest
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Martigues
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Reims
  - Novartis Investigative Site, Rouen
  - Novartis Investigative Site, Saint-Mandé
  - Novartis Investigative Site, Saint-Priest-en-Jarez
  - Novartis Investigative Site, Toulouse
- Germany (16):
  - Novartis Investigative Site, Langenau, Baden-Wurttemberg
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Würzburg, Bavaria
  - Novartis Investigative Site, Halle, Saxony-Anhalt
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Memmingen
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Potsdam
  - Novartis Investigative Site, Schwerin
- Greece (3):
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Chaïdári
  - Novartis Investigative Site, Thessaloniki
- Novartis Investigative Site, Guatemala City, Guatemala
- Hungary (3):
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Kaposvár
  - Novartis Investigative Site, Pécs
- India (4):
  - Novartis Investigative Site, Mysore, Karnataka
  - Novartis Investigative Site, Nagpur, Maharashtra
  - Novartis Investigative Site, Nashik, Maharashtra
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
- Israel (4):
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Tel Aviv
- Italy (7):
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Cona, FE
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Napoli
- Japan (6):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Kisarazu, Chiba
  - Novartis Investigative Site, Ginowan, Okinawa
  - Novartis Investigative Site, Koshigaya, Saitama
  - Novartis Investigative Site, Itabashi-ku, Tokyo
  - Novartis Investigative Site, Osaka
- Novartis Investigative Site, Saida, Lebanon
- Lithuania (2):
  - Novartis Investigative Site, Kaunas, LTU
  - Novartis Investigative Site, Vilnius
- Malaysia (3):
  - Novartis Investigative Site, Kuala Lumpur, Kuala Lumpur
  - Novartis Investigative Site, George Town, Pulau Pinang
  - Novartis Investigative Site, Johor Bahru
- Mexico (2):
  - Novartis Investigative Site, Guadalajara, Jalisco
  - Novartis Investigative Site, Monterrey, Nuevo León
- Novartis Investigative Site, Amersfroort, Utrecht, Netherlands
- Philippines (2):
  - Novartis Investigative Site, Las Piñas
  - Novartis Investigative Site, Makati City
- Poland (5):
  - Novartis Investigative Site, Warsaw, Mazowian
  - Novartis Investigative Site, Ossy
  - Novartis Investigative Site, Rzeszów
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Wroclaw
- Portugal (2):
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Porto
- Russia (6):
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Krasnodar
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Smolensk
  - Novartis Investigative Site, Yaroslavl
- Novartis Investigative Site, Singapore, Singapore
- Slovakia (3):
  - Novartis Investigative Site, Banská Bystrica
  - Novartis Investigative Site, Košice
  - Novartis Investigative Site, Prešov
- South Africa (2):
  - Novartis Investigative Site, Raslouw Centurion, Gauteng
  - Novartis Investigative Site, Soweto, Gauteng
- South Korea (2):
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul
- Spain (10):
  - Novartis Investigative Site, Cadiz, Andalusia
  - Novartis Investigative Site, Granada, Andalusia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Fuenlabrada, Madrid
  - Novartis Investigative Site, Manises, Valencia
  - Novartis Investigative Site, Alicante
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Las Palmas GC
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Pontevedra
- Switzerland (3):
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Geneva
  - Novartis Investigative Site, Lausanne
- Taiwan (2):
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District
- Turkey (Türkiye) (6):
  - Novartis Investigative Site, Aydin, Efeler
  - Novartis Investigative Site, Istanbul, Fatih
  - Novartis Investigative Site, Antalya, Konyaalti
  - Novartis Investigative Site, Kayseri, Melikgazi
  - Novartis Investigative Site, Istanbul, Pendik
  - Novartis Investigative Site, Gaziantep, Sehitkamil
- United Kingdom (8):
  - Novartis Investigative Site, Exeter, Devon
  - Novartis Investigative Site, Dudley, West Midlands
  - Novartis Investigative Site, Bradford, West Yorkshire
  - Novartis Investigative Site, Leeds, West Yorkshire
  - Novartis Investigative Site, Barnsley
  - Novartis Investigative Site, Bristol
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Salford
- Vietnam (2):
  - Novartis Investigative Site, Hanoi
  - Novartis Investigative Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Kimball AB, Bechara FG, Badat A, Giamarellos-Bourboulis EJ, Gottlieb AB, Jemec GBE, Reguiai Z, Villani AP, Alarcon I, Bansal A, Gasperoni F, Martin R, Paguet B, Uhlmann L, Zouater H, Ravichandran S, Alavi A. Long-term efficacy and safety of secukinumab in patients with moderate-to-severe hidradenitis suppurativa: week 104 results from the SUNSHINE and SUNRISE extension trial. Br J Dermatol. 2025 Mar 18;192(4):629-640. doi: 10.1093/bjd/ljae469. PMID 39611771

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study is conducted in 191 centers in 38 countries worldwide
Groups:
- AIN457 Q2WR-Q2W: HiSCR responders at Week 52 who were on Secukinumab every 2 weeks (Q2W) in the core studies and were randomized to Secukinumab Q2W in the Randomized Withdrawal Period (Week 52 to Week 104 or loss of response) in the extension. After loss of response (LOR) or Week 104, patients could continue with open-label Secukinumab 300 mg Q2W
- AIN457 Q2WR-PBO: HiSCR responders at Week 52 who were on Secukinumab every 2 weeks (Q2W) in the core studies and were randomized to placebo in the Randomized Withdrawal Period (Week 52 to Week 104 or loss of response) in the extension. After loss of response (LOR) or Week 104, patients could continue with open-label Secukinumab 300 mg Q2W
- AIN457 Q4WR-Q4W: HiSCR responders at Week 52 who were on Secukinumab every 4 weeks (Q4W) in the core studies and were randomized to Secukinumab Q4W in the Randomized Withdrawal Period (Week 52 to Week 104 or loss of response) in the extension. After loss of response (LOR), patients could continue with open-label Secukinumab 300 mg Q2W. After Week 104, if no LOR, patients could continue with open-label Secukinumab 300 mg Q4W or be up titrated to Q2W at principal investigator discretion.
- AIN457 Q4WR-PBO: HiSCR responders at Week 52 who were on Secukinumab every 4 weeks (Q4W) in the core studies and were randomized to placebo in the Randomized Withdrawal (Week 52 to Week 104 or loss of response) in the extension. After loss of response (LOR) or Week 104, patients could continue with open-label Secukinumab 300 mg Q4W or Q2W at principal investigator discretion
- AIN457 Q2WNR-Q2W: HiSCR non-responders at Week 52 who were on secukinumab every 2 weeks (Q2W) in the core studies and stay on Q2W in the extension
- AIN457 Q4WNR-Q2W: HiSCR non-responders at Week 52 who were on secukinumab every 4 weeks (Q4W) in the core studies and are up-titrated to Q2W in the extension
Period: Overall Study
Arm/Group | AIN457 Q2WR-Q2W | AIN457 Q2WR-PBO | AIN457 Q4WR-Q4W | AIN457 Q4WR-PBO | AIN457 Q2WNR-Q2W | AIN457 Q4WNR-Q2W
Started | 136 | 71 | 121 | 63 | 151 | 157
Full Analysis Set of HiSCR Responders (FAS-R) (All HiSCR responders to whom study treatment was assigned at randomization. Subjects were analyzed according to the treatment assigned to at randomization.) | 136 | 71 | 121 | 63 | 0 | 0
Full Analysis Set of HiSCR Non-responders (FAS-NR) (All HiSCR non-responders to whom study treatment was assigned.) | 0 | 0 | 0 | 0 | 151 | 156
Safety Set (SAF) (All subjects who received at least one dose of study treatment in the extension study. Subjects were analyzed according to the study treatment received.) | 137 | 70 | 121 | 63 | 151 | 156
Completed Randomized Withdrawal Period - Responders Only (This milestone is only applicable to HiSCR responders at Week 52 in the Core studies) | 127 | 64 | 114 | 62 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 136 | 71 | 121 | 63 | 151 | 157
Not completed — Ongoing at the time of the data cut-off date | 94 | 54 | 95 | 43 | 98 | 105
Not completed — Adverse Event | 5 | 3 | 3 | 4 | 6 | 6
Not completed — Lack of Efficacy | 5 | 1 | 3 | 2 | 18 | 7
Not completed — Lost to Follow-up | 5 | 3 | 2 | 2 | 4 | 5
Not completed — Physician Decision | 2 | 0 | 2 | 3 | 1 | 1
Not completed — Pregnancy | 3 | 0 | 3 | 0 | 1 | 2
Not completed — Withdrawal by Subject | 22 | 10 | 12 | 8 | 23 | 31
Not completed — Technical problems | 0 | 0 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AIN457 Q2WR-Q2W | AIN457 Q2WR-PBO | AIN457 Q4WR-Q4W | AIN457 Q4WR-PBO | AIN457 Q2WNR-Q2W | AIN457 Q4WNR-Q2W | Total
Number analyzed (Participants) | 136 | 71 | 121 | 63 | 151 | 157 | 699
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.7 (11.26) | 34.8 (10.55) | 35.4 (12.59) | 36.0 (11.32) | 37.3 (11.00) | 37.1 (11.13) | 36.1 (11.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 38 | 64 | 28 | 91 | 78 | 372
  Male | 63 | 33 | 57 | 35 | 60 | 79 | 327
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 113 | 51 | 90 | 48 | 115 | 111 | 528
  Black or African American | 8 | 6 | 11 | 7 | 6 | 14 | 52
  Asian | 12 | 11 | 13 | 6 | 24 | 28 | 94
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 0 | 1
  American Indian or Alaska Native | 2 | 2 | 5 | 2 | 3 | 3 | 17
  Multiple | 1 | 1 | 2 | 0 | 2 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Time to Loss of Response (LOR) up to Week 104 in Hidradenitis Suppurativa Clinical Response (HiSCR) Responders
Description: Loss of response was defined as:
  * at least a 50% increase in abscess and/or nodules (AN) count compared to the average AN count from the 3 previous visits or at Week 52, whichever is lower and the increase was at least of 3 AN.
  * at least a 30% increase in AN compared to the average AN count from the 3 previous visits or Week 52, whichever is lower, with an increase of at least 2 AN and a further increase in the AN count of at least 2 AN at a re-assessment visit within 2-4 weeks
Time Frame: Up to 52 weeks: from randomization at the extension study (Week 52) up to Week 104 or loss of response. Study day is defined with respect to the core studies.
Population: Full Analysis Set of HiSCR responders (FAS-R)
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | AIN457 Q2WR-Q2W | AIN457 Q2WR-PBO | AIN457 Q4WR-Q4W | AIN457 Q4WR-PBO | AIN457 Q2WNR-Q2W | AIN457 Q4WNR-Q2W
Number analyzed (Participants) | 136 | 71 | 121 | 63 | 0 | 0
Days | 283 [176 to NA] — N/A: Not estimable due to insufficient number of participants with events | 239 [120 to NA] — N/A: Not estimable due to insufficient number of participants with events | 365 [225 to NA] — N/A: Not estimable due to insufficient number of participants with events | 171 [113 to 337] |  |
Statistical Analysis 1: Comparison: AIN457 Q2WR-Q2W vs AIN457 Q2WR-PBO; Test type: Other; p = 0.250, Log Rank; one-sided stratified log-rank test, with region and body weight (<90 kg, ≥ 90 kg) as strata; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.59 to 1.29]
Statistical Analysis 2: Comparison: AIN457 Q4WR-Q4W vs AIN457 Q4WR-PBO; Test type: Other; p = 0.044, Log Rank; one-sided stratified log-rank test, with region and body weight (<90 kg, ≥ 90 kg) as strata; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.47 to 1.05]

2. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: To assess the long-term safety and tolerability of Secukinumab in subjects with moderate to severe hidradenitis suppurativa (HS)
Time Frame: Up to 216 weeks: from randomization at the extension study (Week 52) up to Week 268. Study day is defined with respect to the core studies.
Reporting Status: Not Posted, anticipated posting 2027-07

3. Primary Outcome: Incidence Rate of Participants Achieving Loss of Response (LOR) up to Week 104 in Hidradenitis Suppurativa Clinical Response (HiSCR) Responders
Description: The incidence rate of participants achieving Loss of Response (LOR) was based on the primary estimand.
  * Day 1 = Date of 1st dose intake in the extension study.
  * Subjects at risk = Subjects who did not have LOR and were not censored before or at the start of the specified time interval.
  * Incidence rate (%) = (number of subjects with LOR / number of subjects at risk) x 100.
Time Frame: as for outcome 1
Population: Full Analysis Set of HiSCR responders (FAS-R) with an available value for the outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | AIN457 Q2WR-Q2W | AIN457 Q2WR-PBO | AIN457 Q4WR-Q4W | AIN457 Q4WR-PBO | AIN457 Q2WNR-Q2W | AIN457 Q4WNR-Q2W
Number analyzed (Participants) | 136 | 71 | 121 | 63 | 0 | 0
Percentage of participants
  Day 1 | 0.0 | 0.0 | 0.0 | 0.0 |  |
  2 to 85 days: number analyzed (Participants) | 134 | 71 | 120 | 63 | 0 | 0
  2 to 85 days | 26.9 | 23.9 | 24.2 | 30.2 |  |
  86 to 141 days: number analyzed (Participants) | 97 | 52 | 89 | 43 | 0 | 0
  86 to 141 days | 12.4 | 21.2 | 12.4 | 25.6 |  |
  142 to 197 days: number analyzed (Participants) | 83 | 41 | 76 | 32 | 0 | 0
  142 to 197 days | 8.4 | 9.8 | 6.6 | 9.4 |  |
  198 to 253 days: number analyzed (Participants) | 74 | 37 | 69 | 29 | 0 | 0
  198 to 253 days | 8.1 | 8.1 | 10.1 | 13.8 |  |
  254 to 309 days: number analyzed (Participants) | 67 | 33 | 62 | 25 | 0 | 0
  254 to 309 days | 10.4 | 18.2 | 6.5 | 4.0 |  |
  310 to 351 days: number analyzed (Participants) | 60 | 26.0 | 57 | 24 | 0 | 0
  310 to 351 days | 3.3 | 0.0 | 1.8 | 4.2 |  |
  352 to 399 days: number analyzed (Participants) | 56 | 26 | 56 | 22 | 0 | 0
  352 to 399 days | 5.4 | 0.0 | 5.4 | 9.1 |  |

ADVERSE EVENTS:
Time Frame: From first dose of study treatment in the extension (Week 52) up to the cut-off date for the interim analysis (26-May-2023), approximately 3 years. Study day is defined with respect to the core studies.
Description: Any sign or symptom that occurred during the Randomized Withdrawal Period (for HiSCR responders only) and for the entire study period (from Week 52 up to the cut- off date for the Week 104 interim analysis) for both HiSCR responders and non- responders. The safety analysis were done on the safety population, which included all subjects who received at least one dose of study medication.
Groups:
- Any AIN457 Q4W: All subjects that have been exposed to secukinumab every 4 weeks (Q4W) in the extension study
- Any AIN457 Q2W: All subjects that have been exposed to secukinumab every 2 weeks (Q2W) in the extension study, regardless of responder status at Week 52, including those who up-titrated
- Any AIN457: All subjects exposed to Secukinumab in the extension study regardless of the assigned drug regimen, and regardless of responder status
- AIN457 NR: All subjects who are HiSCR non-responders
Arm/Group | AIN457 Q2WR-Q2W | AIN457 Q2WR-PBO | AIN457 Q4WR-Q4W | AIN457 Q4WR-PBO | Any AIN457 Q4W | Any AIN457 Q2W | Any AIN457 | AIN457 NR
All-Cause Mortality (participants affected / at risk) | 0/137 | 0/70 | 0/121 | 0/63 | 0/180 | 0/637 | 0/687 | 0/307
Serious Adverse Events (participants affected / at risk) | 2/137 | 4/70 | 5/121 | 5/63 | 11/180 | 72/637 | 80/687 | 37/307
Other Adverse Events (participants affected / at risk) | 44/137 | 23/70 | 46/121 | 16/63 | 71/180 | 379/637 | 428/687 | 199/307
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 Q2WR-Q2W (N=137) | AIN457 Q2WR-PBO (N=70) | AIN457 Q4WR-Q4W (N=121) | AIN457 Q4WR-PBO (N=63) | Any AIN457 Q4W (N=180) | Any AIN457 Q2W (N=637) | Any AIN457 (N=687) | AIN457 NR (N=307)
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Keratitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Abdominal adhesions (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Inflammatory bowel disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Intussusception (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Strangulated umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Swollen tongue (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Tongue coated (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 2 | 3 | 2
Breast abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
COVID-19 (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 1
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 3 | 4 | 0
Chronic sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Dermatitis infected (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1
Groin abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Meningitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Sweat gland infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Skin scar contracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Fibrosis tendinous (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Colloid brain cyst (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Optic perineuritis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Schizophrenia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Labia enlarged (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Perineal induration (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Uterine prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Aorto-bronchial fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 1 | 23 | 23 | 14
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Peripheral artery stenosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 Q2WR-Q2W (N=137) | AIN457 Q2WR-PBO (N=70) | AIN457 Q4WR-Q4W (N=121) | AIN457 Q4WR-PBO (N=63) | Any AIN457 Q4W (N=180) | Any AIN457 Q2W (N=637) | Any AIN457 (N=687) | AIN457 NR (N=307)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 8 | 9 | 8
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 4 | 17 | 21 | 10
Toothache (Gastrointestinal disorders) | 1 | 2 | 2 | 0 | 3 | 15 | 18 | 7
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 2 | 6 | 8 | 4
Fatigue (General disorders) | 2 | 0 | 2 | 0 | 2 | 14 | 16 | 6
Pyrexia (General disorders) | 3 | 3 | 1 | 1 | 6 | 21 | 27 | 10
Body tinea (Infections and infestations) | 3 | 0 | 0 | 0 | 0 | 6 | 6 | 1
Bronchitis (Infections and infestations) | 2 | 0 | 0 | 2 | 1 | 28 | 29 | 14
COVID-19 (Infections and infestations) | 11 | 6 | 11 | 7 | 19 | 128 | 147 | 58
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 11 | 11 | 9
Ear infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 13 | 13 | 7
Folliculitis (Infections and infestations) | 0 | 2 | 3 | 2 | 4 | 8 | 12 | 6
Gastroenteritis (Infections and infestations) | 3 | 0 | 2 | 0 | 3 | 11 | 14 | 4
Influenza (Infections and infestations) | 2 | 1 | 2 | 0 | 4 | 22 | 25 | 10
Nasopharyngitis (Infections and infestations) | 5 | 2 | 6 | 2 | 8 | 55 | 63 | 32
Pharyngitis (Infections and infestations) | 0 | 0 | 3 | 0 | 4 | 10 | 14 | 5
Sinusitis (Infections and infestations) | 1 | 0 | 1 | 0 | 4 | 17 | 21 | 9
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 3 | 14 | 17 | 11
Sweat gland infection (Infections and infestations) | 4 | 1 | 1 | 1 | 1 | 14 | 14 | 5
Tonsillitis (Infections and infestations) | 2 | 1 | 0 | 0 | 1 | 15 | 16 | 6
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 3 | 1 | 5 | 28 | 33 | 14
Urinary tract infection (Infections and infestations) | 3 | 2 | 2 | 1 | 3 | 18 | 21 | 7
Alanine aminotransferase increased (Investigations) | 0 | 2 | 0 | 0 | 1 | 7 | 8 | 3
C-reactive protein increased (Investigations) | 1 | 0 | 0 | 0 | 2 | 20 | 22 | 15
SARS-CoV-2 test positive (Investigations) | 0 | 2 | 4 | 2 | 5 | 17 | 22 | 11
Diabetes mellitus (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0 | 0 | 6 | 6 | 2
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0 | 6 | 15 | 20 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 1 | 19 | 20 | 9
Headache (Nervous system disorders) | 3 | 0 | 4 | 0 | 9 | 32 | 41 | 15
Anxiety (Psychiatric disorders) | 0 | 0 | 4 | 0 | 4 | 10 | 14 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0 | 3 | 20 | 23 | 14
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 0 | 1 | 11 | 12 | 6
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0 | 2 | 20 | 22 | 14
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 10 | 11 | 7
Eczema (Skin and subcutaneous tissue disorders) | 3 | 4 | 3 | 1 | 4 | 22 | 26 | 13
Hidradenitis (Skin and subcutaneous tissue disorders) | 6 | 4 | 4 | 3 | 6 | 70 | 75 | 45
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 4 | 0 | 4 | 18 | 22 | 13
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 1 | 14 | 15 | 8
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 17 | 18 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-05-28): https://cdn.clinicaltrials.gov/large-docs/75/NCT04179175/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-22): https://cdn.clinicaltrials.gov/large-docs/75/NCT04179175/SAP_001.pdf